CLINICAL TRIAL: NCT01109160
Title: A Prospective, Open-label Study of Azithromycin for Lymphocytic Bronchiolitis/Bronchitis After Lung Transplantation
Brief Title: Study of Azithromycin for Lymphocytic Bronchiolitis/Bronchitis After Lung Transplantation
Acronym: AZI002
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Principal Investigator, GM. Verleden, Medical Director Leuven Lung Transplant Programme, KU Leuven
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZI002; 2010-018724-16 (EudraCT Number)
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Lymphocytic Bronchi(Oli)Tis Post-lung Transplantation
Keywords: azithromycin; lymphocytic bronchitis or bronchiolitis; lung transplantation; acute allograft rejection; chronic allograft rejection; bronchiolitis obliterans syndrome
MeSH Terms: conditions — Bronchiolitis; Bronchiolitis Obliterans Syndrome | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azithromycin (Experimental): Add-on of study-drug (azithromycin) to 'standard of care': 250 mg daily for 5 days, followed by 250 mg every other day until the end of the study-period (6 months treatment).
  Interventions: Drug: Azithromycin Dihydrate

INTERVENTIONS:
Drug: Azithromycin Dihydrate — Add-on of study-drug (azithromycin) to 'standard of care' at diagnosis of lymphocytic bronchi(oli)tis.
  Study-drug regime: 250 mg daily for 5 days, followed by 250 mg every other day until the end of the study-period (6 months treatment).
  Other Names: Azithromycin 250 mg, ZTM250, Zitromax TM (ATC J01FA10)

SUMMARY:
This study investigates the role of azithromycin treatment for lymphocytic bronchitis/bronchiolitis after lung transplantation.

DETAILED DESCRIPTION:
Lymphocytic bronchitis/bronchiolitis is one of the major risk factors for development of chronic rejection/BOS after lung transplantation. There is currently no established treatment available for this condition. There is now mounting evidence that IL-17 producing lymphocytes (TH17) not only participate in chronic allograft rejection/BOS, but are also present within the airway wall during lymphocytic bronchiolitis and that IL-17 mRNA-levels in bronchoalveolar lavage fluid of these patients are upregulated. As such, TH17 may account for the increased BAL neutrophilia seen in these patients, as IL-17 may be responsible for driving IL-8 secretion (a neutrophil-attracting chemokine) from various cell types in the airways. Since azithromycin has previously been shown to reduce both IL-17 induced IL-8 production by human airway smooth muscle cells 'in vitro' and bronchoalveolar IL-8/neutrophil levels in LTx recipients with established BOS, we believe that azithromycin has great potential for treating lymphocytic bronchi(oli)tis by attenuating this TH17/IL-17/IL-8-mediated airway inflammation, possibly even halting the subsequent development of chronic rejection/BOS after lung transplantation. In this study, histologic, spirometric, bronchoalveolar an radiologic features will be investigated in patients treated with confirmed lymphocytic bronchitis/bronchiolitis treated with azithromycin.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Adult (age at least 18 years old at moment of transplantation)
* Able to take oral medication
* Histologic diagnosis of lymphocytic bronchiolitis or bronchitis ('grade B') without concurrent acute cellular allograft rejection 'grade A' ≥2

Exclusion Criteria:

* Severe suture problems (e.g. airway stenosis) requiring lasering or stenting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-04; Primary Completion 2012-10 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Histology on bronchial and/or transbronchial biopsies | after 3 months of treatment
  Evolution of lymphocytic airway inflammation after 3 months of treatment
Pulmonary function (FEV1) | after 3 months of treatment
  Evolution of FEV1 after 3 months of treatment
Bronchoalveolar cellularity and protein levels (IL-8, IL-17) | after 3 months of treatment
  Evolution of bronchoalveolar cellularity and protein levels (IL-8, IL-17) after 3 months of treatment
Radiologic features | after 3 months of treatment
  Evolution of radiologic features (e.g. tree-in-bud, consolidation, bronchiectasis, air trapping, etc.) on chest X-ray or HRCT after 3 months of treatment

SECONDARY OUTCOMES:
Pulmonary function (FEV1) | after 6 months of treatment
  Evolution of FEV1 after 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Geert M Verleden, MD, PhD, Principal Investigator — KULeuven and UZ Leuven
Locations (1):
- University Hospital Gasthuisberg, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Vanaudenaerde BM, De Vleeschauwer SI, Vos R, Meyts I, Bullens DM, Reynders V, Wuyts WA, Van Raemdonck DE, Dupont LJ, Verleden GM. The role of the IL23/IL17 axis in bronchiolitis obliterans syndrome after lung transplantation. Am J Transplant. 2008 Sep;8(9):1911-20. doi: 10.1111/j.1600-6143.2008.02321.x. PMID 18786233
- [Background] Vanaudenaerde BM, Wuyts WA, Geudens N, Dupont LJ, Schoofs K, Smeets S, Van Raemdonck DE, Verleden GM. Macrolides inhibit IL17-induced IL8 and 8-isoprostane release from human airway smooth muscle cells. Am J Transplant. 2007 Jan;7(1):76-82. doi: 10.1111/j.1600-6143.2006.01586.x. Epub 2006 Oct 25. PMID 17061983
- [Background] Vanaudenaerde BM, Dupont LJ, Wuyts WA, Verbeken EK, Meyts I, Bullens DM, Dilissen E, Luyts L, Van Raemdonck DE, Verleden GM. The role of interleukin-17 during acute rejection after lung transplantation. Eur Respir J. 2006 Apr;27(4):779-87. doi: 10.1183/09031936.06.00019405. PMID 16585086
- [Background] Verleden GM, Vanaudenaerde BM, Dupont LJ, Van Raemdonck DE. Azithromycin reduces airway neutrophilia and interleukin-8 in patients with bronchiolitis obliterans syndrome. Am J Respir Crit Care Med. 2006 Sep 1;174(5):566-70. doi: 10.1164/rccm.200601-071OC. Epub 2006 Jun 1. PMID 16741151